CLINICAL TRIAL: NCT07010614
Title: Theta Burst Modulation of Hippocampal-Cortical Rhythms in Schizophrenia
Brief Title: Brain Stimulation to the Hippocampus in Schizophrenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ethan Andrew Solomon, Postdoctoral Scholar, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 340902
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia Disorders; Mental Disorder; Psychotic Disorder
Keywords: schizophrenia; transcranial magnetic stimulation; TMS; EEG
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- TBS via direct electrical stimulation (Active Comparator): Intracranial electrodes will be used for the delivery of invasive electrical brain stimulation in a theta burst (TBS) pattern.
  Interventions: Device: Intracranial electrodes
- TBS via transcranial magnetic stimulation (Active Comparator): TMS will be used for the delivery of noninvasive brain stimulation in a theta burst (TBS) pattern.
  Interventions: Device: TMS
- Sham TBS via direct electrical stimulation (Sham Comparator): Intracranial electrodes will be used for the delivery of sham invasive brain stimulation (time periods where electrical current is paused).
  Interventions: Device: Intracranial electrodes
- Sham TBS via transcranial magnetic stimulation (Sham Comparator): TMS will be used for the delivery of sham noninvasive brain stimulation (active side of coil turned away from the brain).
  Interventions: Device: TMS sham

INTERVENTIONS:
Device: Intracranial electrodes — Intracranial electrodes will be used for the delivery of invasive electrical brain stimulation.
  Arms: Sham TBS via direct electrical stimulation; TBS via direct electrical stimulation
Device: TMS — TMS will be used for the delivery of noninvasive brain stimulation
  Arms: TBS via transcranial magnetic stimulation
Device: TMS sham — Sham TMS will be used as a comparator for noninvasive brain stimulation
  Arms: Sham TBS via transcranial magnetic stimulation

SUMMARY:
Schizophrenia - marked by delusions, hallucinations, and cognitive deficits - causes the most disability of any mental health condition, but existing treatments have significant side effect burden and are often ineffective. Disordered neural activity in the hippocampus likely contributes to schizophrenia symptoms, but to develop better therapies we need to understand whether hippocampal activity in schizophrenia can be systematically affected by non-invasive brain stimulation techniques like transcranial magnetic stimulation (TMS). This proposal will investigate the use of connectivity-guided theta burst brain stimulation to specifically target hippocampal function in schizophrenia, offering insights into fundamental hippocampal processes, schizophrenia pathophysiology, and potential avenues to use brain stimulation as a therapeutic tool in this devastating illness.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18 to 65 years
* Medically intractable epilepsy requiring phase II monitoring (intracranial EEG arms only)
* DSM-V diagnosis of schizophrenia spectrum Axis I disorders including delusional disorder, brief psychotic disorder, schizophreniform disorder, schizophrenia, schizoaffective disorder (non-invasive TMS-EEG arms only).
* Must have intellectual capacity to ensure adequate comprehension of the study and potential risks involved in order to provide informed consent
* No current or history of major neurological disorders other than epilepsy.

Exclusion Criteria:

* DSM5 diagnosis of intellectual disability
* Significant head injury
* Active suicidal ideation or history of suicide attempt within the past 1 year.
* Medical illness affecting brain structure or function, or other uncontrolled or unstable medical condition.
* Pregnancy or postpartum (<6 weeks after delivery or miscarriage)
* Inability to provide informed consent
* Active substance abuse other than alcohol or cannabis within the past 1 year
* Psychotic illness with a temporal relation to substance use or head injury
* Those with a contraindication for MRIs or TMS (e.g. implanted metal).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in intracranial EEG after one TBS session | 45 minutes
  Change in spontaneous oscillatory EEG power from before to after application of one TBS session, for active and sham stimulation, as measured via intracranial recording electrodes (iEEG).
Change in scalp EEG after one TBS session | 45 minutes
  Change in spontaneous oscillatory EEG power from before to after application of one TBS session, for active and sham stimulation, as measured via scalp recording electrodes (scalp electroencephalography).

SECONDARY OUTCOMES:
Change in TMS-provoked EEG power | 45 minutes
  Change in oscillatory EEG power as provoked by repeated single pulses of TMS, compared from before to after a single session of TBS.
Change in electrical stimulation provoked iEEG power | 45 minutes
  Change in oscillatory iEEG power as provoked by repeated single pulses of invasive electrical stimulation, compared from before to after a single session of TBS.

CONTACTS AND LOCATIONS:
Overall Officials: Ethan A Solomon, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified raw EEG and iEEG data will be shared.
Supporting Information: Analytic Code
Time Frame: Following publication of the data with no end date.
Access Criteria: Anyone who wishes to access the data.